CLINICAL TRIAL: NCT02902640
Title: A Pilot, Multicentric and Observational Study of Safety of Sulfamethoxazole + Trimethoprim + Guaifenesin (Balsamic Bactrim) in Adult Patients With Acute Bronchitis
Brief Title: A Non-Interventional Safety Study of Balsamic Bactrim
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30018
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Bronchitis
MeSH Terms: conditions — Bronchitis | interventions — Guaifenesin; Sulfamethoxazole; Trimethoprim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Acute Bronchitis Participants: Participants with acute bronchitis for whom the treating physician has decided to initiate treatment with Balsamic Bactrim, will be observed. Administration of Balsamic Bactrim will be according to physician's recommendation under local labeling. The study protocol does not enforce any treatment.
  Interventions: Drug: Guaifenesin; Drug: Sulfamethoxazole; Drug: Trimethoprim

INTERVENTIONS:
Drug: Guaifenesin — Guaifenesin will be administered as per treating physician's discretion, according to local labeling. The protocol does not specify any dose, frequency, and duration of treatment.
Drug: Sulfamethoxazole — Sulfamethoxazole will be administered as per treating physician's discretion, according to local labeling. The protocol does not specify any dose, frequency, and duration of treatment.
Drug: Trimethoprim — Trimethoprim will be administered as per treating physician's discretion, according to local labeling. The protocol does not specify any dose, frequency, and duration of treatment.

SUMMARY:
This is a pilot, observational and multicentric study of safety of sulfamethoxazole + trimethoprim + guaifenesin (Balsamic Bactrim) in adult participants with acute bronchitis. Adult participants with acute bronchitis eligible for treatment with Balsamic Bactrim will be enrolled. Administration of Balsamic Bactrim will be according to physician's recommendation under local labeling.

ELIGIBILITY:
Inclusion Criteria:

* Participants starting treatment with Balsamic Bactrim as per treating physician's discretion
* Participants with a clinical diagnosis of acute bronchitis (cough with or without sputum production less than 30 days) according to the treating physician's judgment

Exclusion Criteria:

* Participants who have started treatment with another antibiotic at the time of the visit
* Participants with no respiratory infections
* Participants with mental disorders that do not permit the clinical evaluation of the participant according to the treating physician's criteria
* Participants with severe hepatic parenchymal damage
* Participants with severe renal failure making it difficult to monitor drug plasma concentration
* Participants with hypersensitivity to any of Balsamic Bactrim active ingredients, excipients, and/or sulfas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants receiving treatment for acute bronchitis with Balsamic Bactrim according to standard of care and in line with the current summary of product characteristics (SPC) / local labeling and who have no contraindication to Balsamic Bactrim as per the local label.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events Related to Balsamic Bactrim as Assessed by the Treating Physician | From Day 1 up to end of observation (up to 10 days)

SECONDARY OUTCOMES:
Percentage of Participants With Balsamic Bactrim Dose Change (Increase or Decrease) | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Dose Change by Reason for Change | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Change in Balsamic Bactrim Frequency of Administration | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Dose Interruption | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Treatment Discontinuation | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Balsamic Bactrim Treatment Reintroduction After Discontinuation | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Compliance to Balsamic Bactrim Treatment According to Local Label, as Assessed by Treating Physician | From Day 1 up to end of observation (up to 10 days)
Percentage of Participants With Predisposing Factors (Categories) for Safety (No specific pre-defined factors, these will be decided based on observations during study) | From Day 1 up to end of observation (up to 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Peru (4):
  - Clínica Providencia; Centro de Investigación de Enfermedades Respiratorias, Lima
  - Clinica de Especialidades Medicas, Lima
  - Clinica San Borja; Instituto de Enfermedades Respiratorias EFEH, Lima
  - Centro de Investigaciones Medicas/Hospital Maria Auxiliadora, San Juán de Miraflores

REFERENCES:
- [Derived] Falcon M, Iberico C, Guerra F, Reyes I, Felix E, Flores M, de Los Rios J, Diaz ME, Casas A, Sanchez-Gambetta S, Carrasco R. A pilot study of safety of sulfamethoxazole, trimethoprim and guaifenesin in pediatric and adult patients with acute bronchitis. BMC Res Notes. 2019 Mar 4;12(1):119. doi: 10.1186/s13104-019-4150-2. PMID 30832720